CLINICAL TRIAL: NCT00522886
Title: Determination of the Toxicity of Standard Dose Cetuximab Together With Concurrent Individualised, Isotoxic Accelerated Radiotherapy and Cisplatin-vinorelbine for Patients With Stage III Non-small Cell Lung Cancer: A Phase I Study
Brief Title: Phase I Cetuximab and Concurrent Radio-chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Academisch Ziekenhuis Maastricht (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Prof. Dr. Dirk De Ruysscher, Maastricht Radiation Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-03-009
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: cetuximab; concurrent; iso-toxic; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cetuximab — Eligible patients will be given 2 cycles(of 21 days) of carboplatin (AUC 5) day 1 and gemcitabine (1250 mg/m2) days 1,8. Patients without progressive disease will be entered in the phase I dose-escalation part of the study. Chest radiation will be given concurrently with cetuximab, cisplatin and vinorelbine, which will be escalated in 3 steps until dose-limiting toxicity occurs.
  14 days after the last gemcitabine (=day 43), radiotherapy is started : First 3 weeks: 1.5 Gy BID to a dose of 45 Gy in 30 fractions, then 2 Gy QD to a mean lung dose of 19 Gy. Cetuximab: 400 mg/m2 7 days before radiotherapy (= day 36) and during the course of radiotherapy a weekly dose 250 mg/m2. Cetuximab will be delivered at the same days as chemotherapy.
  Cisplatin(all steps): 50 mg/m2 days 43, 50; 40 mg/m2 day 64.
  Vinorelbine:
  Step 1: 10 mg/ m2 days 43, 50; 8 mg/m2 days 66 and 73. Step 2: 20 mg/ m2 days 43, 50; 8 mg/m2 days 66 and 73. Step 3: 20 mg/ m2 days 43, 50; 15 mg/m2 days 66 and 73.

SUMMARY:
To determine the MTD toxicity of standard dose cetuximab together with concurrent individualized, isotoxic accelerated radiotherapy and cisplatin-vinorelbine

DETAILED DESCRIPTION:
Phase I trial with escalating doses of vinorelbine and standard doses of radiotherapy, cisplatin and cetuximab.

Eligible patients receive 2 cycles of carboplatin (AUC 5) day 1 and gemcitabine (1250 mg/m2) days 1,8. One cycle duration is 21 days.

Patients without progressive disease (PD) according to the RECIST criteria (appendix 1) will be entered in the phase I dose-escalation part of the study. Chest radiation is given concurrently with cetuximab, cisplatin and vinorelbine. The latter drug will be escalated in three steps until dose-limiting toxicity occurs.

On day 43, i.e. 14 days after the last gemcitabine delivery, radiotherapy is started.

Radiotherapy: In all patients in every dose-step, the radiation will be given as follows: first 3 weeks: 1.5 Gy BID to a dose of 45 Gy in 30 fractions, then 2 Gy QD to a mean lung dose (MLD, this is related to radiation-induced lung damage) of 19 Gy. Maximum dose: 69 Gy given in 5.5 weeks. Maximum dose to the spinal cord: 50 Gy.

Cetuximab: All patients will receive a starting dose 400 mg/ m2 7 days before the beginning of radiotherapy (i.e. day 36), thereafter a weekly dose 250 mg/ m2 during the course of radiotherapy for 5 consecutive weeks. Cetuximab will be delivered at the same days as chemotherapy.

Cisplatin: In all patients in every dose-step, cisplatin will be given as follows: Step 1, 2 and 3: 50 mg/ m2 days 43, 50; 40 mg/m2 day 64.

Vinorelbine will be escalated in three steps:

Step 1: 10 mg/ m2 days 43, 50; 8 mg/m2 days 66 and 73. Step 2: 20 mg/ m2 days 43, 50; 8 mg/m2 days 66 and 73. Step 3: 20 mg/ m2 days 43, 50; 15 mg/m2 days 66 and 73.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer
* Inoperable stage III (UICC 2002; sixth edition) (no pleural effusion)
* WHO performance status 0 or 1
* Less than 10% weight loss in the last 6 months
* Lung function: FEV1 at least 50% and DLCO at least 50% of the predicted value
* No recent severe cardiac disease
* Adequate bone marrow function
* Adequate renal function
* Adequate hepatic function
* Life expectancy more than 6 months
* Measurable cancer
* Willing and able to comply with study prescriptions
* 18 years or older
* Not pregnant or breast feeding
* Written informed consent
* No previous radiotherapy to the chest

Exclusion Criteria:

* Not non-small cell lung cancer histology
* Mixed pathology
* History of prior chest radiotherapy
* Recent (<3 months) myocardial infarction
* Uncontrolled infectious disease
* Less than 18 years old
* Inadequate pulmonary function
* Other active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) 3 months after the ende of chemo-radiation | 3 months

SECONDARY OUTCOMES:
During and after chemo-radiation: (CTC 3.0) Dysphagia, Cough, Dyspnea, Skin rash, Myelitis, Neuropathy, Neutrophiles, Platelets, Hemoglobin, Diarrhea, Renal failure, Liver dysfunction, Tumour response 3 m. after end chemo-radiation and Survival | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD PhD, Principal Investigator — Maastro Clinic, The Netherlands; Anne-Marie Dingemans, MD PhD, Principal Investigator — academisch ziekenhuis Maastricht, azM
Locations (1):
- Maastricht Radiation Oncology, MAASTRO clinic, Maastricht, Limburg, Netherlands